CLINICAL TRIAL: NCT00990171
Title: The Effects Nutrition Status and Body Composition On Peritoneal Dialysis Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200906084R
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Peritoneal Dialysis; Wasting and Malnutrition
Keywords: peritoneal Dialysis; wasting and malnutrition; nutrition status; bioelectrical impedance analysis; body composition
MeSH Terms: conditions — Cachexia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma dianeal
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PD-BCM: 1. Patients at National Taiwan University Hospital (NTUH)
  2. Patients who have received PD more than 3 months
  3. Patients who sign the informed consents
  4. Patients who aged between 20-90 years

SUMMARY:
A prospective long-term follow up of peritoneal dialysis patients' outcome correlates with nutritional status and body composition.

DETAILED DESCRIPTION:
Wasting and malnutrition are common and serious complications in patients on peritoneal dialysis and are strongly associated with adverse outcomes. Techniques for assessing nutrition have limitations and, due to metabolic effects and confounding effects of altered hydration and other body composition abnormalities, these limitations are greater in the context of renal failure. Bioelectrical impedance analysis is a promising method for the objective assessment and monitoring of body composition. Body composition techniques subdivide the body into compartments on the basis of differing physical properties. The different compartments reflect hydration, nutrition/wasting, body fat, and bone mineral content, which are all of great importance in patients on peritoneal dialysis. We will conduct a prospective long-term follow up of PD patients' outcome correlates with nutritional status and body compositions. The patients will receive BIA every three months, and other routine clinical data such as dialysis adequacy, peritoneal equilibration test and monthly biochemical data are collected to analyze. An additional blood sample 8 ml and 5 ml dialysate of overnight, 0 hour, 2 hour and 4 hour will be collected during annual PET for other inflammatory cytokines and nutritional markers such as adiponectin, leptin, ghrelin, prealbumin and transferrin. The follow up period will be as long as possible and the last recruited into this study is in the Aug 2014. These data will be used for the morbidity and mortality analysis to see if body compositions will be more useful and timely than the other nutritional parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at National Taiwan University Hospital
2. Patients who have received PD more than 3 months
3. Patients who sign the informed consents

Exclusion Criteria:

1. Patients who have received PD less than 3 months
2. Patients who refuse to sign informed consents
3. Patients who refuse to draw additional blood for research

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Measure BCM could be a nutrition status marker | 5 yrs

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan